CLINICAL TRIAL: NCT03600259
Title: Cohort Study of Acute Myocardial Infarction in Tianjin
Brief Title: Tianjin Inpatient Acute Myocardial Infarction Registry
Acronym: TAMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tianjin Chest Hospital (Other)
Responsible Party: Principal Investigator, Yin Liu,MD, Director, Cardiology Department, Tianjin Chest Hospital, Tianjin Chest Hospital
Other Study IDs: TAMI20180705
Record Dates: First submitted 2018-07-06; First posted 2018-07-26 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Infarction, Acute
Keywords: Myocardial Infarction; Coronary Disease; Coronary Artery Disease; Myocardial Ischemia
MeSH Terms: conditions — Myocardial Infarction; Coronary Disease; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Myocardial Infarction

SUMMARY:
Acute myocardial infarction(AMI) is the most serious manifestation of coronary artery disease. AMI is characterized by high mortality, high disability, and high cost. However, multicenter research on AMI with large sample size in Tianjin or even China is limited. By including AMI in 36 hospitals,this multicenter study will capture the changes in epidemiological trends ,analyze the status of treatment in Tianjin, and explore the best treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with acute myocardial infarction according to Cardiac biomarker values [Selective cardiac troponin (cTc) elevation and/or decline detection, at least one value exceeds the 99% reference limit (URL) and at least one of the following:（1）Symptoms of myocardial ischemia；（2）New or suspected new obvious ST-T changes or new left bundle branch block (LBBB)；（3）ECG pathological Q waves；（4）Image evidence of recent loss of viable myocardium, or new regional wall motion abnormalities；（5）Coronary thrombosis confirmed by angiography or autopsy.]

Exclusion Criteria:

* Those who did not meet the diagnosis of acute myocardial infarction (no myocardial ischemia-related symptoms, elevation of markers of myocardial necrosis and imaging findings of myocardial infarction); those who met the inclusion criteria but refused to participate in the study; The researchers judged that the subjects had poor compliance and could not Complete follow-up as required.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with acute myocardial infarction from 36 hospitals in Tianjin were enrolled between January 2015 and January 2020
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac death | 1 year
  Due to recent cardiac causes (eg myocardial infarction, low-volume heart failure, fatal arrhythmias), any deaths from unknown and unexplained deaths and all surgical-related deaths (including treatment-related deaths) will be attributed to cardiac death.Unless there is a clear non-cardiological cause, all deaths are considered heart disease. Specifically, even patients with concurrent potentially fatal non-cardiac diseases (such as cancer, infections) who have any accidental death should be classified as having a heart attack.

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 10 days on average (during hospitalization)
  Composite of major adverse cardiovascular events (MACE) including cardiac death, heart failure, target vessel revascularization, recurrent myocardial infarction, stroke, severe bleeding
Major adverse cardiovascular events | 1 month
  Composite of major adverse cardiovascular events (MACE) including cardiac death, heart failure, target vessel revascularization, recurrent myocardial infarction, stroke, severe bleeding
Major adverse cardiovascular events | 3 months
  Composite of major adverse cardiovascular events (MACE) including cardiac death, heart failure, target vessel revascularization, recurrent myocardial infarction, stroke, severe bleeding
Major adverse cardiovascular events | 6 months
  Composite of major adverse cardiovascular events (MACE) including cardiac death, heart failure, target vessel revascularization, recurrent myocardial infarction, stroke, severe bleeding
Major adverse cardiovascular events | 1 year
  Composite of major adverse cardiovascular events (MACE) including cardiac death, heart failure, target vessel revascularization, recurrent myocardial infarction, stroke, severe bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Yin Liu, M.D, Principal Investigator — Tianjin Chest Hospital
Locations (1):
- Tianjin Chest Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gao MD, Zhang EY, Liu YY, Li XW, Xiao JY, Sun GY, Liu Y. Intracoronary pressure gradient measurement in acute myocardial infarction patients with the no-reflow phenomenon during primary percutaneous coronary intervention. Chin Med J (Engl). 2020 Apr 5;133(7):766-772. doi: 10.1097/CM9.0000000000000709. PMID 32149760